CLINICAL TRIAL: NCT02203240
Title: Dietary Cocoa for Inhibition of Metabolic Endotoxemia and Glucose Intolerance
Brief Title: Cocoa and Metabolic Health in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: The Hershey Company (Industry)
Responsible Party: Principal Investigator, Andrew P. Neilson, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VT13261005
Record Dates: First submitted 2014-07-26; First posted 2014-07-29 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Prediabetes
Keywords: Cacao; Polyphenols; Prediabetic State; Blood Glucose; Glucose Intolerance; Diabetes Mellitus, Type 2; Obesity; Muscle, Skeletal; Endotoxins; Gut Permeability; Incretins; Metabolic Flexibility
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Diabetes Mellitus, Type 2; Obesity | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cocoa (Experimental): 3 servings of polyphenol-rich cocoa beverage consumed per day.
  Interventions: Other: Cocoa
- Placebo (Placebo Comparator): 3 servings of non-cocoa beverage consumed per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Cocoa
  Arms: Cocoa
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the impact of consuming cocoa on blood glucose levels, glucose metabolism, and other markers of pre-diabetes in overweight and/or obese individuals. Our hypothesis is that consumption of cocoa improves insulin sensitivity and glucose metabolism in subjects at risk for developing type-2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than or equal to 25 and less than 40.
* Have at least one of the following: 1) impaired fasting glucose (IFG) after an overnight fast with plasma glucose concentration between 100-125 mg/dl, 2) impaired glucose tolerance (IGT) as identified by the standard Oral Glucose Tolerance Test (OGTT) with 2 hour plasma glucose concentration between 140-200 mg/dl following 75 g glucose OGTT, 3) HbA1c levels between 5.7-6.4% or 4) considered at risk to developing type 2 diabetes by the American Diabetes Association risk assessment. If subjects are above the prediabetic range for any of these tests (indicating they may be type 2 diabetic), they will be excluded and referred to their physician.
* Weight stable (+/-2 kg) for the last 6 months.
* Sedentary to recreationally active (less than 2 d/wk, 20 min/d).
* Have a blood pressure that is less than 160/100 mmHg, total cholesterol that is less than 300 mg/dl and a triglyceride concentration of less than 450 mg/dl.

Exclusion Criteria:

* Past or current history of coronary heart disease, stroke or major cardiovascular disease events, respiratory diseases, endocrine or metabolic diseases (including type 1 and type 2 diabetes), inflammatory bowel disease, cancer, or neurological or hematological disorders that would compromise the study or the health of the subject.
* Past or current history of gastrointestinal disorders (including lactose intolerance, ulcers, cancer (stomach, intestinal, colon, pancreatic, liver, etc) NASH, NAFLD, cirrhosis, IBD/IBS, celiac disease, etc).
* Current use of any medication including but not limited to cholesterol lowering medication (including fibric acid derivatives and niacin), antibiotics, immunosuppressive drugs, azole antifungals, non-steroidal anti-inflammatory drugs (NSAIDs), hormone replacement therapy or antioxidants/supplements.
* Use of antibiotics, prebiotics, or probiotics within the prior 3 months.
* Smoking or other tobacco use
* Habitual consumption of alcohol more than 2 servings/d for males and 1 serving/d for females.
* Strict vegetarians or vegans, or strong aversions to major food groups that may be part of the controlled diet.
* Recent surgery
* History of alcohol or drug abuse.
* Pregnant or plan to become pregnant
* Allergic to either lidocaine or bupivacaine

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Baseline and 4 weeks
  Insulin sensitivity will be determined using Bergman's minimal model (MINMOD Millennium software) via a frequently sampled intravenous glucose tolerance test (IVGTT). Fasting baseline blood samples will be taken prior to the dextrose injection (0.3 g/kg; 50% solution) at minute 0. Venous samples will be collected at minutes 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, and 18. Insulin (0.025 U/kg) will be injected at minute 20. Venous sampling will continue at minutes 22, 23, 24, 25, 27, 30, 40, 50, 60, 70, 80, 90, 100, 120, 150, and 180. Glucose concentration will be immediately analyzed an automated glucose oxidase analyzer. Insulin will be later measured from serum using the Immulite 1000 immunoassay analyzer.

SECONDARY OUTCOMES:
Change in blood glucose response to a mixed meal | Baseline and 1 week
  The test meal will be 2-8 oz. servings of a meal replacement beverage providing a mixed macronutrient profile, supplemented with either a cocoa beverage dry mix (10 g cocoa) or a calorie-matched placebo beverage mix (0 g cocoa). Blood samples will be taken at baseline and subsequently 1, 2, 3, and 4 hours after the first sip of the test beverage. Plasma glucose concentrations will be analyzed immediately using a glucose auto-analyzer (Yellow Springs Instruments).
Change in hormone secretion response to a mixed meal | Baseline and 1 week
  Serum insulin, GLP-1, GIP, and C-peptide concentrations will be determined using commercially available enzyme-linked immunosorbent assay (ELISA) kits from the blood samples drawn at baseline, 1, 2, 3, and 4 hours during the mixed meal challenge.
Change in skeletal muscle metabolic flexibility | Baseline and 4 weeks
  Subjects will consume a high fat meal containing 820 kcal; 52 g total carbohydrates, 24 g protein, and 58 g fat. During the high fat challenge session, two skeletal muscle biopsies will be conducted on alternate legs; one before the high fat meal and one 4 hours later. Biopsies of the vastus lateralis will be performed using a 5 mm modified Bergström needle. Collected tissue will be washed in 0.9% sterile saline to remove blood and tissue. Samples will be weighed and added to buffer and placed on ice for immediate analysis of substrate flexibility. For substrate flexibility, pyruvate oxidation will be used to assess the activity of pyruvate dehydrogenase. Calculated metabolic flexibility is expressed as a ratio of pyruvate oxidation to pyruvate oxidation + free fatty acids.
Change in blood endotoxin levels | Baseline and 4 weeks
  During the high fat challenge (see Outcome 4), blood samples will be collected at baseline and 1, 2, 3, and 4 h after the first bite of the meal. Serum endotoxin will be measured in duplicate using Limulus Amebocyte Lysate Pyrogent ® 5000 assay kits.
Change in gut permeability | Baseline and 4 weeks
  The four-sugar [40 g sucrose, 1 g mannitol, 1 g sucralose and 5 g lactulose] probe test will be used to assess total gut permeability. After an overnight fast and urine evacuation, participants will be asked to consume the sugar-probe beverage within 5 minutes. They will be given two breakfast sandwiches to consume immediately. Participants will be instructed to collect all of their urine in a provided container from the time the beverage was consumed (0 h) until 5 h. A second urine collection container will be filled between 6-24 h. Twenty-four hours later, the volume of urine in each container will be measured and aliquots collected for later analysis. Gastroduodenal permeability is defined as sucrose/mannitol ratio (0-5 h). Small intestinal permeability is defined as the calculated lactulose/mannitol ratio for 0-5 samples. Colonic permeability is defined as both the 6-24 h lactulose/mannitol ratio and 6-24 h sucralose/mannitol ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Neilson, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Human Integrative Physiology Laboratory, Blacksburg, Virginia, United States